CLINICAL TRIAL: NCT05018858
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Lupus
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for Lupus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-20-ATG-4
Record Dates: First submitted 2021-08-20; First posted 2021-08-24 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Lupus
Keywords: Lupus; Lupus Arthritis; stem cell treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Lupus

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Lupus. This patient funded trial aims to study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of Lupus. Patients with Lupus will receive a single intravenous infusion of UC-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease an autologous T-Cell vaccine will be utilized created from the patient's own cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lupus
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Athens Beverly Hills Medical Group, Glyfada, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Li J, Zhang Y, Zhang M, Chen J, Li X, Hu X, Jiang S, Shi S, Sun L. Umbilical cord mesenchymal stem cell transplantation in active and refractory systemic lupus erythematosus: a multicenter clinical study. Arthritis Res Ther. 2014 Mar 25;16(2):R79. doi: 10.1186/ar4520. PMID 24661633
- [Background] Wang D, Zhang H, Liang J, Li X, Feng X, Wang H, Hua B, Liu B, Lu L, Gilkeson GS, Silver RM, Chen W, Shi S, Sun L. Allogeneic mesenchymal stem cell transplantation in severe and refractory systemic lupus erythematosus: 4 years of experience. Cell Transplant. 2013;22(12):2267-77. doi: 10.3727/096368911X582769c. PMID 24388428
- [Background] Sun L, Wang D, Liang J, Zhang H, Feng X, Wang H, Hua B, Liu B, Ye S, Hu X, Xu W, Zeng X, Hou Y, Gilkeson GS, Silver RM, Lu L, Shi S. Umbilical cord mesenchymal stem cell transplantation in severe and refractory systemic lupus erythematosus. Arthritis Rheum. 2010 Aug;62(8):2467-75. doi: 10.1002/art.27548. PMID 20506343